CLINICAL TRIAL: NCT04776330
Title: Study Evaluating Safety and Efficacy of BCMA-Targeted Prime CAR-T Cell in Patients With Relapsed/Refractory Multiple Myeloma and Plasma Cell Disease
Brief Title: a Clinical Research of BCMA-Targeted Prime CAR-T Cell Therapy in Relapsed/Refractory Multiple Myeloma and Plasma Cell Disease
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chongqing Precision Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PBC027
Record Dates: First submitted 2021-02-26; First posted 2021-03-01 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Multiple Myeloma; Neoplasm, Plasma Cell; Multiple Myeloma in Relapse
Keywords: Multiple Myeloma; BCMA; prime Chimeric Antigen Receptor T Cell
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BCMA targeted prime CAR-T cells treat (Experimental): Patients will be be treated with BCMA targeted prime CAR-T cells
  Interventions: Biological: BCMA targeted prime CAR-T cells

INTERVENTIONS:
Biological: BCMA targeted prime CAR-T cells — BCMA targeted prime CAR-T cell therapy

SUMMARY:
This is a single arm study to evaluate the efficacy and safety of BCMA-targeted prime CAR-T cells therapy for patients with relapsed/refractory Multiple Myeloma.

DETAILED DESCRIPTION:
There are limited options for treatment of relapse/refractory Multiple Myeloma. BCMA is expressed on most Multiple Myeloma cells so it is an ideal target for CAR-T. In this study, investigators will evaluate the safety and efficacy of prime CAR- T targeting BCMA in patients with relapsed/refractory Multiple Myeloma. The primary goal is safety and efficiency assessment, including adverse events and disease status after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent;
2. Diagnose as relapsed /refractory multiple myeloma or other plasma cell disease, and meet one of the following conditions:

   1. Failed to standard chemotherapy regimens;
   2. Relapse after complete remission, high-risk and / or refractory patients ;
   3. Relapse after hematopoietic stem cell transplantation;
3. Evidence for cell membrane BCMA expression
4. All genders, ages: 18 to 75 years#
5. The expect time of survive is above 3 months;
6. KPS>60
7. No serious mental disorders ;
8. Left ventricular ejection fraction ≥50%
9. Sufficient hepatic function defined by ALT/AST≤3 x ULN and bilirubin≤2 x ULN;
10. Sufficient renal function defined by creatinine clearance≤2 x ULN;
11. Sufficient pulmonary function defined by indoor oxygen saturation≥92%; 12. With single or venous blood collection standards, and no other cell collection contraindications;

13. Ability and willingness to adhere to the study visit schedule and all protocol requirements.

Exclusion Criteria:

1. Previous history of other malignancy;
2. Presence of uncontrolled active infection;
3. Evidence of disorder that need the treatment by glucocorticoids;
4. Active or chronic GVHD
5. The patients treatment by inhibitor of T cell
6. Pregnant or breasting-feeding women;
7. Any situation that investigators regard not suitable for attending in this study (e.g. HIV , HCVinfection or intravenous drug addiction) or may affect the data analysis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-03-07 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Adverse events that related to treatment | 2 years
  Therapy-related adverse events will be recorded and assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0)
The response rate of BCMA targeted prime CAR-T treatment in patients with relapse/refractory Multiple Myeloma that treatment by BCMA targeted prime CAR-T cells therapy | 2 years
  The response rate of BCMA targeted prime CAR-T treatment will be recorded and assessed according to the IMWG

SECONDARY OUTCOMES:
Rate of BCMA targeted prime CAR-T cells in bone marrow and peripheral blood | 2 years
  In vivo (bone marrow and peripheral blood) rate of BCMA targeted prime CAR-T cells were determined by means of flow cytometry
Quantity of BCMA targeted prime CAR copies in bone marrow and peripheral blood | 2 years
  In vivo (bone marrow and peripheral blood) quantity of BCMA targeted prime CAR copies were determined by means of qPCR
Quantity of clonal plasma cells in bone marrow | 1 years
  In vivo (bone marrow) quantity of clonal plasma cells
Levels of IL-6 in Serum | 1years
  In vivo (Serum) quantity of IL-6
Duration of Response (DOR) of BCMA targeted prime CAR-T treatment in patients with refractory/relapsed multiple myeloma | 2 years
  DOR will be assessed from the first assessment of sCR/CR/VGPR/PR to the first assessment of recurrence or progression of the disease or death from any cause (censored)
Progress-free survival(PFS) of BCMA targeted prime CAR-T treatment in patients with refractory/relapsed multiple myeloma | 2 years
  PFS will be assessed from the first prime CAR-T cell infusion to death from any cause or the first assessment of progression (censored)
Overall survival(OS) of BCMA targeted prime CAR-T treatment in patients with refractory/relapsed multiple myeloma | 2 years
  OS will be assessed from the first prime CAR-T cell infusion to death from any cause (censored)

CONTACTS AND LOCATIONS:
Overall Officials: Sanbin Wang, MD, Principal Investigator — 920th Hospital of Joint Logistics Support Force of People's Liberation Army of China; Cheng Qian, PhD, Principal Investigator — Chongqing University Cancer Hospital
Locations (1):
- 920th Hospital of Joint Logistics Support Force, Kunming, Yunnan, China